CLINICAL TRIAL: NCT01148368
Title: A Clinical Trial to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety of Fimasartan in Renal Impairment Patients and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A657-BR-CT-113
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2010-12

CONDITIONS: Renal Impairment
Keywords: fimasartan; renal impairment; hypertension
MeSH Terms: conditions — Renal Insufficiency; Hypertension | interventions — fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal impairment patients (Experimental): renal impairment patients who eGFR is lower than 30 ml/min/1.73m^2 without hemodialysis
  Interventions: Drug: fimasartan
- healthy volunteers (Active Comparator): healthy volunteers group
  Interventions: Drug: fimasartan

INTERVENTIONS:
Drug: fimasartan — single administration of fimasartan 120mg

SUMMARY:
The purpose of this study is to compare and evaluate the pharmacokinetic characteristics and the safety of fimasartan in renal impairment patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

<Renal impairment patient>

* age: 20-65 years
* eGFR: < 30ml/min/1.73m^2
* not on dialysis
* body weight: greater than 55kg
* written informed consent

<Healthy volunteer>

* age: 20-65 years
* body weight: greater than 55kg
* written informed consent

Exclusion Criteria:

* AST, ALT > 1.5 times of upper normal range
* positive drug or alcohol screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic characteristic of fimasartan | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 32, 48h
  AUC, Cmax, Tmax, T1/2, and CL/F of fimasartan

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea